CLINICAL TRIAL: NCT03545555
Title: Investigations on the Effect of Kale on the Lipid Status (Untersuchungen Zum Einfluss Von Grünkohl Auf Den Lipidstatus)
Brief Title: Investigations on the Effect of Kale on the Lipid Status
Acronym: HypocholKale
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Jena (Other)
Responsible Party: Principal Investigator, Volker Boehm, Head of Bioactive Plant Products Research Group, University of Jena
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: AGBAP2018-1
Record Dates: First submitted 2018-05-07; First posted 2018-06-04 (Actual); Last update posted 2018-06-04 (Actual); Status verified 2018-05

CONDITIONS: Effects of Kale Ingredients on Lipid Status Parameter
Keywords: kale; antioxidant capacity; cholesterol; lipid status

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Kale Powder (Experimental): 5 capsules with kale preparation "kale powder" per day for 8 weeks
  Interventions: Dietary Supplement: Kale Preparation "Kale Powder"
- Kale Extract (Experimental): 5 capsules with kale preparation "kale extract" per day for 8 weeks
  Interventions: Dietary Supplement: Kale Preparation "Kale Extract"
- Flavonoid Extract (Experimental): 5 capsules with kale preparation "flavonoid extract" (from kale) per day for 8 weeks
  Interventions: Dietary Supplement: Kale Preparation "Flavonoid Extract"
- Placebo (Placebo Comparator): 5 capsules with "placebo" per day for 8 weeks
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Kale Preparation "Kale Powder" — Effect of kale preparation kale powder on lipid status
  Arms: Kale Powder
Dietary Supplement: Kale Preparation "Kale Extract" — Effect of kale preparation kale extract on lipid status
  Arms: Kale Extract
Dietary Supplement: Kale Preparation "Flavonoid Extract" — Effect of kale preparation flavonoid extract on lipid status
  Arms: Flavonoid Extract
Dietary Supplement: Placebo — Effect of placebo on lipid status
  Arms: Placebo

SUMMARY:
This intervention study investigates the effects of various kale preparations (dietary supplements) on lipid status parameters. Within the study period of 8 weeks, three blood withdrawals are planned (week 0, 4 and 8) for the volunteers. Lipid status parameters (total cholesterol, HDL cholesterol, LDL cholesterol, triacylglycerides) will be determined in blood. There is a correlation between contents of LDL cholesterol, total cholesterol and triacylglycerides and the risk for cardiovascular diseases (CVD). In contrast, a high content of HDL cholesterol is correlated with a lower risk for CVD. In addition, the contents of apolipoprotein A1 and apolipoprotein B will be analysed.

ELIGIBILITY:
Inclusion Criteria:

* total cholesterol > 200 mg/dl

Exclusion Criteria:

* LDL cholesterol < 130 mg/dl
* medication to lower blood lipids
* genetically based hypercholesterolemia

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2018-04-13 (Actual); Primary Completion 2018-09 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Change of lipid status parameters | weeks 0, 4 and 8
  total cholesterol, HDL cholesterol, LDL cholesterol

SECONDARY OUTCOMES:
Change of apolipoproteins | weeks 0, 4 and 8
  apolipoprotein A1 and apolipoprotein B
Change of antioxidant capacity | weeks 0, 4 and 8
  lipophilic antioxidant capacity (L-TEAC)

CONTACTS AND LOCATIONS:
Locations (1):
- Friedrich Schiller University, Institute iof Nutritional Science, Jena, Thuringia, Germany